CLINICAL TRIAL: NCT06042504
Title: Effects of Family Status of Osteopathic Medical Students on Their Perceived Level of Stress.
Status: Completed | Type: Observational
Sponsor: The Touro College and University System (Other)
Responsible Party: Principal Investigator, Tommaso Meregalli, Principal Investigator, The Touro College and University System
Other Study IDs: 2206E
Record Dates: First submitted 2023-09-09; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Married students with no children: Submit Survey
  Interventions: Other: Survey
- Married students with children: Submit Survey
  Interventions: Other: Survey
- Unmarried Students with children: Submit Survey
  Interventions: Other: Survey
- Familial caregiver: Submit Survey
  Interventions: Other: Survey
- Unmarried without kids: Submit Survey
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Subjects will complete a survey. The survey consists of two parts, "A" and "B". During part "A" subjects will indicate which of the 5 cohorts they identify as. Successively in part "B", subject will complete a survey known as the "Perceived Stress Scale" (PSS).

SUMMARY:
The investigators are interested in studying the effects of familial obligations, including marriage, parenthood, familial caregiving, on stress levels in Osteopathic Medical Students (OMS). The investigators expect to find that having a family may increase the stress level of OMS in comparison with OMS who don't have familial obligations.

ELIGIBILITY:
Inclusion Criteria:

* Medical Students

Exclusion Criteria:

* Not current Medical Students

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, female, other
Study Population: Current Medical Students
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2023-09-09 (Actual)

PRIMARY OUTCOMES:
Total PSS Score | Through study completion, an average of 1 year.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Touro College of Osteopathic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No